CLINICAL TRIAL: NCT00833404
Title: Effects of Smoking Cessation on Sexual Health in Men
Brief Title: Smoking Cessation and Sexual Health in Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Christopher Harte, Ph.D., Postdoctoral fellow, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-06-0020
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: Smoking Cessation
Keywords: Smoking; Smoking Cessation; Quit Smoking; Stop Smoking; Nicotine Patch; Nicotine Replacement Therapy; Sexual Functioning; Erectile Functioning; Sexual Health
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smoking Cessation (Experimental): 8-week nicotine patch regimen
  Interventions: Drug: Nicotine transdermal patch
- Wait List Control (No Intervention): Smoking as usual

INTERVENTIONS:
Drug: Nicotine transdermal patch — 8-week nicotine patch regimen (21mg/day during week 1-4, 14mg/day during week 5-6, and 7mg/day during week 7-8).
  Other Names: Nicotine; Nicotine patch
  Arms: Smoking Cessation

SUMMARY:
This is a 12-week clinical trial investigating the effects of smoking cessation on sexual functioning in men. This study consists of 3 sessions and provides 8 weeks of free nicotine transdermal patches. It is hypothesized that men who quit smoking, compared to men who smoke as usual, will demonstrate improved sexual functioning, measured both physiologically (erectile functioning) and subjectively (self-reported sexual functioning).

DETAILED DESCRIPTION:
Objective: Tobacco use constitutes the single most preventable cause of disease and death in the world today and is responsible for introducing a number of diseases including many types of cancer, cardiovascular diseases, and respiratory diseases. Extensive literature indicates that cigarette smoking is an independent risk factor for introducing erectile impairment in men. Controlled clinical trials examining the effects of smoking cessation on sexual functioning are necessary in order to investigate whether quitting smoking improves sexual health.

Design: This is a 12-week clinical trial in which 80 male long-term smokers will be tested at baseline (while smoking) and then randomized to an 8-week nicotine patch treatment regimen (n = 50) or to a delayed treatment wait list condition (n = 30). All participants will be reassessed at mid-treatment (4 weeks), and at 1-month follow-up.

Main Outcome Measures: Physiological (penile circumferential change via penile plethysmography), and subjective (continuous self-report) sexual responses to erotic stimuli will be examined, as well as global changes in self-reported sexual functioning.

Implications: If participants do in fact demonstrate a significant increase in sexual arousal and sexual functioning as a result of smoking cessation, these results may have the potential for facilitating programs and interventions targeting the prevention and cessation of cigarette smoking in men. This would alleviate enormous economic burdens caused by erectile dysfunction and other smoking-related diseases.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Between the ages of 25 and 60
* Proficient in English
* Currently smoke at least 15 cigarettes per day for at least 5 years
* Heterosexual
* Currently sexually active (sexual intercourse within the past 30 days)
* Committed to quit smoking

Exclusion Criteria:

* History of HIV infection or active, untreated pelvic or urinary tract infection including, sexually transmitted diseases such as chlamydia genital herpes, gonorrhea, or syphilis.
* Major pelvic surgery that may have caused nerve damage, or serious bladder, rectal, or abdominal surgery.
* Neurological impairment due to diabetes, stroke, pelvic nerve damage secondary to trauma, cancer treatments, myasthenia gravis, multiple sclerosis or spinal cord damage.
* Clinically significant untreated renal or endocrine disease.
* Uncontrolled hypotension or hypertension manifested by systolic blood pressure >170 or <90 mm Hg or diastolic blood pressure >100 or <50 mm Hg.
* History of serious drug abuse or serious alcohol abuse within the past 12 months (>= 16 points on the Alcohol Use Disorders Identification Test (AUDIT) and >= 6 on the Drug Abuse Screening Test (DAST-10).
* Evidence of schizophrenia, bipolar disorder, delusional disorder, or psychotic disorders not classified elsewhere as per the DSM-IV
* Using medications known to affect sexual or vascular functioning, including antidepressants and anti-hypertensives, as well as sildenafil, vardenafil, tadalafil, or any other substance designed to affect sexual performance
* Patients using insulin, narcotic pain relievers (propoxyphene, pentazocine), tricyclic antidepressants, oxazepam, or medications for respiratory diseases such as COPD or asthma (xanthines (e.g., theophylline) as these drugs are contraindicated by the nicotine patch
* Patients who report experiencing clinically significant sexual difficulties, including hypoactive sexual desire disorder, sexual arousal disorder, premature ejaculation, or inhibited orgasm prior to the onset of smoking.
* Recent myocardial infarction, serious heart arrhythmias, and those with serious or worsening angina.
* Hypersensitivity or allergy to nicotine.
* History of or current psoriasis, dermatitis (atopic or eczematous), active peptic ulcers, severe renal impairment, hyperthyroidism, pheochromocytoma, or insulin-dependent diabetes mellitus.

Ages: 23 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-01 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Sexual functioning | Baseline, 4 weeks, 12 weeks

SECONDARY OUTCOMES:
Cardiovascular health | Baseline, 4 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christopher B Harte, MA, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States